CLINICAL TRIAL: NCT00689975
Title: The Effects of a Combined Diet and Exercise Intervention on Biomarkers Associated With Disease Recurrence After Breast Cancer Treatment: The Sheffield DEBRA Trial
Brief Title: Diet and Exercise or Normal Care in Overweight or Obese Women Who Have Undergone Treatment for Stage I, Stage II, or Stage III Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Hallam University (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized
Other Study IDs: CDR0000588427; SHU-USMS-DEBRA; ISRCTN08045231; EU-20821
Record Dates: First submitted 2008-06-03; First posted 2008-06-04 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2009-12

CONDITIONS: Breast Cancer
Keywords: stage IA breast cancer; stage IB breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Counseling; Flow Cytometry; Immunoenzyme Techniques

INTERVENTIONS:
Behavioral: behavioral dietary intervention
Behavioral: exercise intervention
Other: counseling intervention
Other: flow cytometry
Other: immunoenzyme technique
Other: laboratory biomarker analysis
Procedure: complementary or alternative medicine procedure
Procedure: standard follow-up care

SUMMARY:
RATIONALE: Studying diet and exercise interventions in overweight and obese patients with breast cancer may help doctors learn more about how to help patients lose weight and change their body composition.

PURPOSE: This randomized clinical trial is studying diet and exercise to see how well it works compared with normal care in overweight or obese women who have undergone treatment for stage I, stage II, or stage III breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To examine the effects of a dietary and exercise intervention on body weight and body composition in overweight or obese women who have undergone breast cancer treatment.
* To examine the effects of a dietary and exercise intervention on indices of psychological health status and biomarkers associated with disease recurrence in overweight or obese women who have undergone breast cancer treatment.

Secondary

* To examine the relationship between change in body weight and biomarkers associated with disease recurrence and physiological health status, including circulating levels of estrogen, C-reactive protein, and interleukin-6.
* To examine the relationship between changes in psychological health status, circulating stress hormones, and indices of immune function.
* To examine the effects of the dietary and exercise intervention on broader quality-of-life dimensions.

OUTLINE: Patients are randomized to one of intervention arms.

* Arm I (lifestyle intervention): Patients undergo moderate-intensity aerobic-exercise sessions 3 to 5 days a week for 24 weeks. Patients not able to attend five supervised sessions are counseled on how they can fit an extra 1-2 home/community-based exercise sessions into their weekly routine. All sessions of physical activity are recorded in a physical activity log. Portable pedometers are used to determine the number of steps/distance walked each day. Patients wear heart-rate monitors throughout the exercise sessions. Heart rate and ratings of perceived exertion are assessed at regular intervals. The exercise-therapy sessions use a variety of cognitive-behavioral techniques for promoting exercise adherence as well as positive attitudes and experiences.

Patients are also given individualized healthy-eating dietary advice and written information packet named ' Weight Loss On A Plate'. Patients are also counseled on how to reduce their dietary fat intake to 25% of total caloric intake, eating at least 5 portions of fruit and vegetables daily, increasing fiber intake, reducing carbohydrates, and taking moderate amounts of alcohol. Patients are also counseled on how to reduce their total daily calorie intake to 600 kcal below their calculated energy requirements. Individual energy requirements will be estimated from a formula of basal metabolic rate and physical activity level. Patients complete a 3-day diet diary prior to beginning study treatment and then weekly throughout the study. The diaries from pre-intervention and from weeks 6, 12, 18, and 24 are analyzed, looking specifically at macronutrients. Patients meet with the research assistant once weekly to discuss their individual diet diaries and identify ways in which they can further improve their nutritional intake.

* Arm II (normal care): Patients are provided with a general healthy-eating booklet entitled, "Getting the Balance Right".

Depression, psychological stress, and quality of life are assessed at baseline and then at 12 weeks, and 25 weeks.

Blood samples are examined for various biomarkers including interleukin-6 by ELISA, estradiol by radioimmunoassay, and for lymphocyte phenotyping and NK-cell activity by flow cytometry.

Salivary cortisol levels are measured 4 times on two consecutive days by high-sensitivity salivary cortisol enzyme immunoassay.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of stage I, II, or III breast cancer

  * No metastatic breast cancer
  * No inoperable or active loco-regional disease
* Body mass index (BMI) > 25
* Patients must have completed treatment for breast cancer within the past 3-18 months
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Female
* Menopausal status not specified
* Willing and able to attend supervised exercise sessions at least 3 times per week for a period of 24 weeks
* Patients must be an exercise pre-contemplator, contemplator, or preparer as defined by the transtheoretical model
* No physical/psychiatric impairment that would seriously impair physical mobility
* No severe nausea, anorexia, or other diseases affecting health (e.g., arthritis and multiple sclerosis)
* More than 3 months since prior exercise and not currently engaged in exercise (two or more times per week for at least 30 minutes per session)

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Concurrent tamoxifen, other endocrine treatments, and trastuzumab (Herceptin®) allowed
* No concurrent alternative/complementary diets
* No concurrent high-dose antioxidant supplement therapy
* More than 4 months since prior and no concurrent hormone-replacement therapy or oral contraceptives

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2006-02; Primary Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Body weight
Body composition

SECONDARY OUTCOMES:
Pychological stress via the Perceived Stress Scale
Depression via the Beck Depression Inventory II
Cardiorespiratory fitness
Quality of life via the FACT-G and FACT-B

CONTACTS AND LOCATIONS:
Overall Officials: John M. Saxton, PhD, Principal Investigator — Royal Hallamshire Hospital
Locations (1):
- Sheffield Hallam University - City Campus, Sheffield, England, United Kingdom

REFERENCES:
- [Result] Saxton JM, Daley A, Woodroofe N, Coleman R, Powers H, Mutrie N, Siddall V, Crank H. Study protocol to investigate the effect of a lifestyle intervention on body weight, psychological health status and risk factors associated with disease recurrence in women recovering from breast cancer treatment [ISRCTN08045231]. BMC Cancer. 2006 Feb 9;6:35. doi: 10.1186/1471-2407-6-35. PMID 16469108